CLINICAL TRIAL: NCT03700450
Title: Cyclophosphamide as Graft-versus-host Prophylaxis After Allogeneic Stem Cell Transplantation for Multiple Myeloma. A Phase II Study (Allo-MM-PostCy-Study)
Brief Title: Cyclophosphamide as Graft-versus-host Prophylaxis After Allogeneic Stem Cell Transplantation for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Esteve Pharmaceuticals GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Allo-MM-PostCy-Study
Record Dates: First submitted 2018-08-23; First posted 2018-10-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Without detection of deletion 17p or translocation 4;14;; Post Cyclophosphamide; GvHD Prophylaxis; Allogeneic SCT
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: All patients will receive on day 3 and 4 after allogeneic stem cell transplantation 50 mg/kg BW cyclophosphamide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclophosphamid post Tranplant (Experimental): Patients will receive on day 3 and 4 after allogeneic stem cell transplantation 50 mg/kg BW cyclophosphamide
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Patients will receive on day 3 and 4 after allogeneic stem cell transplantation 50 mg/kg BW cyclophosphamide
  Other Names: Endoxan

SUMMARY:
The present study is a multicenter, prospective phase II-study to evaluate the chronic GvHD and progression-free survival at 2 years after after allogeneic stem cell transplantation for patients with multiple myeloma.

DETAILED DESCRIPTION:
The present study is a multicenter, prospective Phase II-study to evaluate the incidence of acute and chronic graft-versus-host disease at 2-years, the 2-year risk of non-relapse mortality, the 2-year progressive-free, and overall survival in patients with multiple myeloma who received a toxicity-reduced conditioning regimen combined of thiotepa and busulfan followed by allogeneic stem cell transplantation from matched or mismatched, related/unrelated and haploidentical donor, and cyclophosphamide as post-transplant GvHD prophylaxis in comparision to a historical group.

In this study will further determine toxicity and safety of cyclophosphamide as GvHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma newly diagnosed with deletion 17p or translocation 4;14 or multiple myeloma with 1. or 2. relapse after autologous stem cell transplantation
2. Patients age: 18 - 65 years at time of inclusion (female and male)
3. Performance status ECOG < 2
4. Availability of haploidentical, matched or mismatched related or unrelated donor
5. Patients understand and voluntarily sign an informed consent
6. The study population includes female of childbearing potential (FOCP). FOCP have to agree to comply with the applicable contraceptive requirements of the protocol as named below for the duration of the study and 6 months after end of study or having post-menopausal status or be permanently sterilized (at least 6 weeks post-sterilization).
7. Men who are sexually active with FOCP must be instructed to use male contraception (condom) in order to avoid exposure of an existing embryo/fetus. Contraception should be continued until 6 months after end of study.

Exclusion Criteria:

1. Severe active infection or other uncontrolled severe conditioning
2. Severe renal, hepatic, pulmonary or cardiac disease, such as:

   * Total bilirubin, SGPT or SGOT > 3 times upper the normal level
   * Left ventricular ejection fraction < 30 %
   * Creatinine clearance < 30 ml/min
   * DLCO < 35 % and/or receiving supplementary continuous oxygen
3. Positive serology for HIV
4. Pregnant or lactating women (positive serum pregnancy test)
5. Women of child-bearing potential with unclear contraception
6. Age < 18 and > 65 years.
7. Uncontrolled invasive fungal infection at time of screening (baseline)
8. Serious psychiatric or psychological disorders
9. Participation in another study with ongoing use of unlicensed investigational product from 28 days before study enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Chronic GvHD | 2 years
  Chronic GvHD at 2 years after allogeneic SCT
Progression-free survival | 2 years
  Progression-free survival at 2 years after allogeneic SCT

SECONDARY OUTCOMES:
Non-relapsed mortality | 2 years
  Non-relapsed mortality at 2 years after allogeneic SCT
Acute GvHD | Day +100 after allogeneic SCT
  Incidence of acute GvHD on Day +100 after allogeneic SCT
Chronic GvHD | 1 and 2 years after allogeneic SCT
  Incidence of chronic GvHD at 1 and 2 years after allogeneic SCT
Toxicity of cyclophosphamide | till 2 years
  Toxicity scored according to NCI CTCAE, Version 4.0
Remission rate | till 2 years
  Complete remission rate (including sCR and MRD negativity)
Overall Survival | 2 years
  Overall survival at 2 years
Progression-free Survival | 2 years
  Progression-free survival at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kröger, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (3):
- Germany (3):
  - University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz

IPD SHARING:
Plan to Share IPD: No